CLINICAL TRIAL: NCT04425278
Title: Study of tDCS Intervention on Motivational Anhedonia of Major Depressive Disorder
Brief Title: tDCS Intervention on Motivational Anhedonia of Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Fengqiong Yu, A/Prof., Anhui Medical University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Yu
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Transcranial Direct Current Stimulation; Major Depressive Disorder; Event-Related Potentials
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Real Stimulation (Active Comparator): The Real Stimulation of tDCS lasted 20 mins.Behavior and ERPs dataset should be acquired before the first tDCS session and after the last tDCS session.
  Interventions: Device: transcranial direct current stimulation with real current
- Sham Stimulation (Sham Comparator): The Sham Stimulation of tDCS lasted 20 minutes with no current. In particular, the current went up for the first 30 seconds and went down for the last 30 seconds.Behavior and ERPs dataset should be acquired before the first tDCS session and after the last tDCS session.
  Interventions: Device: transcranial direct current stimulation with sham current
- Control (No Intervention): Behavior and ERPs dataset should be acquired before and after 14 days.

INTERVENTIONS:
Device: transcranial direct current stimulation with real current — transcranial direct current stimulation with real current is a noninvasive technique to activate and modify the activity of the neurons
  Arms: Real Stimulation
Device: transcranial direct current stimulation with sham current — transcranial direct current stimulation with sham current is a placebo
  Arms: Sham Stimulation

SUMMARY:
Study of tDCS intervention on motivational anhedonia of Major Depressive Disorder

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after transcranial direct current stimulation (tDCS) treatment. Patients were randomly allocated to real group , sham group or control group. A threshold of 3 points on the Hamilton Depression scale has been specified by the National Institute for Health and Care Excellence to determine a clinically meaningful difference between active pharmacotherapy and placebo. We plan to enroll minimum total sample size of 37 participants in real, sham or control group respectively according to the Power and Sample Size program. The decision to enroll a patient was always made prior to randomization. The tDCS administrators had access to the randomization list. They had minimal contact with the patients, and no role in assessing depression. Each patient would be treated for continuous 14 days by tDCS in real and sham group. The control group was evaluated by clinical symptom scale, behavioral evaluation before and after 14 days.

Before the tDCS treatment, depression symptom of each participant was assessed by the Hamilton Depression Scale and the Beck Depression Self-Rating Scale. The anhedonia severity was evaluated by The Temporal Experience of Pleasure Scale, the Self-Report Apathy Evaluation Scale, Dimensional Anhedonia Rating Scale, the Motivation and Pleasure Scale.The neuroimaging data was collected using event-related potentials during monetary incentive delay task. After the last treatment, the same scales and neuroimaging scan were used again to assess the treatment effect of the tDCS and the underlying brain mechanism. Each participant was interviewed in detail about the adverse event of the tDCS intervention during the past 14 days.Every participant should take part in the study in voluntary and sign an informed consent form before the study.

ELIGIBILITY:
Inclusion Criteria:

1. Meet criteria of depression assessed by at least two psychiatrists according to the five version of Diagnostic and Statistical Manual of Mental Disorders.
2. The score of Hamilton Depression Rating Scale-17 was larger than 18.
3. Patients were taking antidepressants--Selective Serotonin Reuptake Inhibitor(SSRIs) alone.
4. Age was between 18 to 60 year old.
5. The education duration was at least 6 years.
6. The vision or corrected vision was normal.
7. Right handedness.
8. No treatment of rTMS, transcranial direct current stimulation or electroconvulsive therapy before.

Exclusion Criteria:

1. History of significant head trauma or neurological disorders.
2. Alcohol or drug abuse.
3. Focal brain lesions.
4. History of seizure.
5. First degree relative with epilepsy, significant neurological illness or head trauma, endocrine disease.
6. Significant unstable medical condition.
7. Recent aggression or other forms of behavioral dyscontrol.
8. Left-handedness.
9. Pregnancy.
10. Current alcohol or drug abuse
11. Inability to provide informed consent.
12. Patients with contraindications or factors affecting imaging quality, such as pacemakers, cochlear implants, or hearts Cerebrovascular metal stent, and metal denture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Hamilton Depression Scale | baseline;14 day post-treatment
  The participants' depression symptom assessed by the Hamilton Depression Scale change from baseline after the treatment.
Change from baseline in Motivation and Pleasure Scale | baseline;14 day post-treatment
  The severity of participants' anhedonia assessed by the Motivation and Pleasure Scale change from baseline after the treatment.

SECONDARY OUTCOMES:
The change from baseline in behavioral results of Monetary Incentive Delay task | baseline; 14 day post-treatment change from baseline after the treatment.
  The motivational anhedonia assessed by accuracy and response time in Monetary Incentive Delay task
The change from baseline in event-related brain potentials during the monetary incentive delay task | baseline; 14 day post-treatment
  The amplitudes of brain potentials of contingent negative variation and P3 assessed by event-related brain potentials methods change from baseline after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, MD, Study Chair — Anhui Medical University; Fengqiong Yu, MD, Study Director — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, Anhui, China